CLINICAL TRIAL: NCT01786928
Title: Impact of Resistance Training During Hospitalization in COPD Patients: a Randomized and Controlled Trial
Brief Title: The Role of Resistance Exercise in Chronic Obstructive Pulmonary Disease Exacerbation
Acronym: RECOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Celso Ricardo Fernandes de Carvalho, PhD in physiology, University of Sao Paulo
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTR-001-RCB
Record Dates: First submitted 2012-01-10; First posted 2013-02-08 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease; exacerbation; resistance training; muscle force
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- resistance training (Experimental): resistance training of the upper and lower limbs, two series of 80% of repetition maximum test
  Interventions: Other: Resistance training
- Control (No Intervention): Traditional Respiratory Therapy for bronchial hygiene

INTERVENTIONS:
Other: Resistance training — Resistance training group received training program for upper (shoulder flexion and abduction and biceps) and lower limbs (knee extension and flexion and hip flexion). Daily exercise for every muscle was performed with free weights at 80% of an maximal repetition test and a 4 minutes rest was allowed between each step.
  Arms: resistance training

SUMMARY:
The purpose of this study is to determine whether resistance exercise are effective in combating the decline in muscle strength during an exacerbation of Chronic Obstructive Pulmonary Disease (COPD).

DETAILED DESCRIPTION:
Acute exacerbations are common in patients with COPD and cause specific signs and symptoms, such as increased dyspnea, productive cough with altered sputum, and fever. With disease progression, exacerbations are frequent and have a negative impact on health related quality of life and pulmonary function as well as increase mortality. More severe exacerbations require hospitalization resulting in enormous health expenditures, severely reducing daily life activities and declining peripheral muscle strength that can be only partially reversed after 3 months. Despite many features have been pointed out as responsible for the decrease in muscle strength during hospitalization, physical inactivity seems the most important.

Resistance training is an interesting therapeutic option to prevent and/or reverse muscular dysfunction due to immobilised in healthy subjects and stable COPD patients because induces hypertrophy of type II fibers, increases muscle strength and exercise tolerance. In addition, provokes lower dyspnea perception during effort compared with other exercise training. Despite these benefits for stable COPD, the impact of a resistance exercise program during hospitalization remains poorly known.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized for exacerbation of COPD

Exclusion Criteria:

* patients presenting change in mental status (confusion, lethargy or coma)
* persistence or worsening in hypoxemia (PaO2<40mmHg) and/or respiratory acidosis (pH<7.25) despite oxygen supplementation or use of non-invasive ventilation
* hemodynamic instability requiring vasoactive drugs
* patients transferred to ICU
* hospitalization lower than 5 days
* diseases that prevented the exercises

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The benefits of resistance training during exacerbation of COPD on peripheral muscle strength during hospitalization | Will be evaluated on the second day of hospitalization, the day of hospital discharge (this time interval must be longer than five days)
  The metric used to evaluate the strength gain is given in kilogram (absolute value) and percentage relative to that obtained on the second hospital day

SECONDARY OUTCOMES:
The benefits of resistance training during exacerbation of COPD on physical activity in daily life | Will be evaluated in the third and fifth day of hospitalization and thirty days after discharge
  The metric used to evaluate the changes will be given in minutes and percentage of total time

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo C Borges, specialist, Study Chair — school of Medicine university of sao paulo
Locations (1):
- University Hospital of sao paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Borges RC, Carvalho CR. Impact of resistance training in chronic obstructive pulmonary disease patients during periods of acute exacerbation. Arch Phys Med Rehabil. 2014 Sep;95(9):1638-45. doi: 10.1016/j.apmr.2014.05.007. Epub 2014 May 28. PMID 24879965